CLINICAL TRIAL: NCT05220228
Title: The Effect of 2mg Sub-acute Prucalopride on Cognition and Emotional Processing in Participants Recovered From Depression
Brief Title: Prucalopride and Cognition in Recovered Depression
Acronym: PROGRESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: R77135/RE001
Record Dates: First submitted 2022-01-25; First posted 2022-02-02 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Depression in Remission
Keywords: Cognition; Emotional processing
MeSH Terms: interventions — prucalopride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prucalopride (Experimental): Prucalopride - 1mg for 2 days, and then increased to 2mg for a further 5-8 days. Testing will occur on day 7 ideally, but may take place up to and including day 10.
  Interventions: Drug: Prucalopride
- Placebo (Placebo Comparator): Placebo (sucrose / lactose) for 7-10 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prucalopride — 1mg prucalopride x 2d, 2mg prucalopride x 5-8d
  Other Names: Resolor; Montegrity; Axunio
  Arms: Prucalopride
Drug: Placebo — Lactose / sucrose placebo
  Arms: Placebo

SUMMARY:
The current study has two aims:

1. To test the effect of 5-HT4 receptor agonism on cognition (including memory, attention and cognitive control) in individuals with previous history of depression.
2. To explore if prucalopride has an effect on emotional processing biases consistent with its effects on serotonin.

DETAILED DESCRIPTION:
Cognitive impairment within depression is common and appears to be at least partly separate from the mood component. It is not well targeted by current treatments and it may persist even after remission of mood symptoms. Therefore, it may be clinically beneficial to search for new therapies that are able to improve cognition in those who have, or are recovering from, depression.

Agonists of the serotonin receptor subtype 4 (5-HT4) have shown two profiles of effect in animal models: (i) a pro-cognitive profile, improving in learning and memory on a range of rodent paradigms; and (ii) an antidepressant-like profile, reducing depression and anxiety-related behaviours in rodent models of depression and anxiety.

A previous study in our group examining acute prucalopride administration (1mg) in 40 healthy human volunteers found improvements in learning and memory but little effect on emotional processing. This pro-cognitive effect was supported by a subsequent study where healthy volunteers received 7 days of prucalopride. In this study, prucalopride led to both better performance on a visual memory task, and increased activation in the hippocampus and an associated memory processing region in response to a memory stimulus. As short-term treatment with clinically-effective antidepressants such as SSRIs is known to produce positive biases in the processing of emotional information in healthy volunteers, this lack of effect on emotional processing was not consistent with prucalopride having antidepressant potential, and is surprising considering the strength of the animal data. One factor that has not yet been explored is whether the translation was limited due to the low dose of prucalopride used in our previous study.

Therefore, we wish to see if we (i) can translate this pro-cognitive effect of prucalopride into participants with a previous history of depression and current mild cognitive issues; and (ii) can use a full treatment dose of prucalopride to evaluate its effect on emotional processing.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the research
* Male or female
* Body mass index in the range of 18 to 33
* Not currently taking any medications (except for contraception), including being antidepressant free for at least three months
* Have at least two previous episodes of depression, and have been recovered from the most recent episode of depression for six months
* Current PHQ-9 score < 10 (the cut off for DSM major depression)

Exclusion Criteria:

The participant may not enter the study if ANY of the following apply:

* Any current Axis 1 DSM-5 psychiatric disorder
* Any previous episode of a severe mental illness, other than Depressive Disorder. Comorbid Anxiety disorders will be allowed, but not OCD (Obsessive Compulsive Disorder) or PTSD.
* A first degree relative diagnosed with Bipolar Affective Disorder Type 1 or Schizophrenia
* Body Mass Index outside the range of 18 to 33 inclusive
* Any significant current medical condition likely to interfere with conduct of the study or analysis of data
* Current use of psychoactive and / or medically significant medication as judged by a study medic, whether prescribed or bought over the counter (the contraceptive pill, the Depo-Provera injection or the progesterone implant will not result in exclusion)
* Ongoing psychopharmacological treatment for depression, including hypnotics (psychotherapy will be allowed as long as not newly-started in the last 6 weeks)
* High consumption of licit substances to an extent that would make complying with study protocol challenging (including alcohol, caffeine, nicotine)
* Past history of dependence to illicit substances, and any consumption of illicit substances in the three months prior to the study
* Currently pregnant or breast feeding
* Current, or a significant history of, gastro-intestinal disorder or irritable bowel syndrome
* Known lactase deficiency or any other problem absorbing lactose, galactose, or glucose
* Participation in a study that involves the use of a medication or novel vaccine within the last three months
* Participation in a study using the same tasks in the last two years
* Any physical (including visual and auditory) or language impairment that would make complying with the study protocol challenging

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
Performance (accuracy) across cognitive battery | Day 7-10
  To investigate the pattern of effects of sub-acute administration of 2mg prucalopride versus placebo on a battery of cognitive measures including attention (DSST), memory (AVLT), executive function (TMT-A/B), working memory (N-back), and reward sensitivity (PILT).

SECONDARY OUTCOMES:
FERT | D7-10
  Accuracy (%) and reaction times on computer-based task of facial expression recognition (FERT), comparing those receiving drug and placebo.
ECAT/EREC/EMEM | D7-10
  Number of positive and negative words correctly categorised, recalled, and recognised on emotional memory task, comparing those receiving drug and placebo.
FDOT | D7-10
  Reaction times to fearful, happy, and neutral faces in masked and unmasked conditions (FDOT), comparing those receiving drug and placebo.
Emotional go/no-go | D7-10
  Reaction time and accuracy, comparing those receiving drug and placebo.
PDQ-20 | D7-10
  Change of score from baseline, comparing those receiving drug and placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Angharad de Cates, MRCPsych, Principal Investigator — University of Oxford
Locations (1):
- Department of Psychiatry, Warneford Hospital, University of Oxford, Oxford, Oxfordshire, United Kingdom